CLINICAL TRIAL: NCT06810258
Title: Diagnostic and PROgnostic BIOmarkers Before and After Kidney Transplantation
Brief Title: BIOmarkers Before and After Kidney Transplantation
Acronym: PROBIOT
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240374
Record Dates: First submitted 2024-12-05; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Kidney Disease; Kidney Transplantation
Keywords: Biomarkers; Chronic kidney disease; Kidney transplantation
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One or two 50 mL urine tubes and 17.5 mL blood tubes are collected. The urine cell pellet is recovered from each sample by centrifugation and lysed according to a well-defined protocol established by the manufacturer and then stored at -80°C.
  * The PaXgen tube is left at room temperature for 2 hours according to the protocol and then stored at -20°C.
  * Serum is recovered after centrifugation of the dry tube at 4000 rpm for 10 minutes and stored at -80°C.
  * PBMC are extracted from the Cpt tube, frozen at 50% in SVF-10% DMSO and stored at -80°C.
  Depending on the study, mRNA expression is then analysed by quantitative PCR (targeted research) or microarray.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sample during native kidney biopsy — blood sample during standard of care visit for a native kidney biopsy (17.5mL)
Other: Blood sample during renal graft biopsy — blood sample during standard of care visit for a renal graft biopsy (17.5mL)
Other: Urine sample during renal graft biopsy — Urine sample during standard of care visit for a renal graft biopsy (50mL)
Other: Urine sample during native kidney biopsy — Urine sample during standard of care visit for a native kidney biopsy (50mL)

SUMMARY:
In clinical nephrology, the search for urinary, blood and tissue biomarkers of specific kidney diseases is an important goal. In recent years, the use of these biomarkers has made it possible to diagnose many renal diseases that affect the native kidney. In some cases, biomarkers may be useful in determining the evolutionary profile of the disease and thus the most appropriate therapeutic management.

DETAILED DESCRIPTION:
In clinical nephrology, the search for urinary, blood and tissue biomarkers of specific kidney diseases is an important goal. In recent years, the use of these biomarkers has made it possible to diagnose many renal diseases that affect the native kidney. In some cases, biomarkers may be useful in determining the evolutionary profile of the disease and thus the most appropriate therapeutic management.

The progression of these kidney diseases sometimes necessitates kidney transplantation for patients undergoing follow-up. Although the one-year survival rate for kidney transplantation has improved significantly over the last decade and is currently 90%, long-term survival is not increasing. Renal graft biopsy remains the reference method for the diagnosis and prognosis of various post-transplant conditions. This method has two limitations: i) it is an invasive procedure associated with complications, which means that it cannot be performed systematically on a large scale throughout the transplant process; ii) the sample size is limited and does not always allow a reliable prognosis to be made. The identification of urinary or blood biomarkers with diagnostic and prognostic value would allow an earlier diagnosis than that made by kidney biopsy. This would allow patients to be treated specifically and individually at an early stage, before damage to the kidney graft occurs, and would significantly improve long-term kidney graft survival.

The main objective of this study is to investigate blood, urine and tissue biomarkers in renal pathologies for diagnostic and prognostic purposes.

As this is an observational study, the main criteria of interest for analysis will include

* Exposure factors: blood and/or urine and/or tissue biomarkers
* Diagnostic criteria (presence or absence of the kidney disease of interest) and prognostic criteria (occurrence or absence of the event of interest).

Once the patient has been informed and has consented to participate in the study, and once the selection criteria have been verified:

1. Clinical data will be recorded in the medical record as part of routine care and then collected in the research database. Clinical data collected will include demographic, biological, clinical and imaging data.
2. The following samples will be collected at one time during the routine care examinations 17.5 mL of additional blood: 1 x 5 mL dry tube, 1 x 10 mL CPT tube and 1 x 2.5 mL PAXgen tube.
3. The excess of urine samples (50 to 100 mL) collected during the course of treatment is retained;
4. If kidney biopsies are performed as part of treatment, part of the sample will be diverted to the biological collection: 1 fragment, 5x5x5 mm.

For patients undergoing native renal biopsy:

A single blood and urine sample (17.5 ml blood: serum, PBMC, RNA) will be collected on the day of the renal biopsy.

In kidney transplant patients:

On the day of the kidney biopsy, patients will be admitted to the day hospital. An additional blood sample (17.5 ml blood: serum, PBMC, RNA) will be taken for each kidney biopsy performed as part of standard care. A urine sample (one to two 50 mL urine tube) is collected.

These blood, urine and tissue samples may be stored in a biological collection and used for constitutional genetic studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalised for renal biopsy of a native kidney or for renal transplantation
* Age >18 years
* Informed and consented
* Covered by a social security scheme

Exclusion criteria:

* Patients under guardianship, conservatorship or legal protection
* Pregnant or breastfeeding
* Patient deprived of liberty
* Patients of legal age who are unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated in the nephrology and transplantation department of Henri Mondor Hospital who have had a biopsy of their native kidneys or renal graft or enlisted in the renal allograft waiting list
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2034-10-08 (Estimated); Study Completion 2035-10-08 (Estimated)

PRIMARY OUTCOMES:
The main aim of this study is to identify blood, urine and tissue biomarkers in kidney disease for diagnostic and prognostic purposes. | 1 year
  the main criteria of interest for the analysis will include :
  * Exposure factors: blood and/or urine and/or tissue biomarkers
  * Diagnostic (presence or absence of the renal disease of interest) and prognostic (occurrence or absence of the event of interest) endpoints

SECONDARY OUTCOMES:
improve understanding of the pathophysiological mechanisms involved in the development of native kidney pathologies | through study completion, an average of 1 year
  These samples may also be used to conduct studies aimed at enhancing the understanding of: the pathophysiological mechanisms involved in the development of native kidney diseases (e.g., acute cellular or humoral rejection, chronic graft dysfunction, BK virus nephropathy, etc.), and factors predictive of tolerance and response to treatment, which could lead to the identification of new therapeutic biomarkers and therapeutic targets.
  The choice of markers is still highly exploratory, but we would mention: CXCL10, CXCL9, FoxP3, Vimentin

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Henri Mondor, Créteil, France